CLINICAL TRIAL: NCT04667624
Title: A Randomized, Open Label, Single Dose, 2-sequence, 4-period, Cross-over Phase I Clinical Trial to Compare and Evaluate the Safety and PK After Oral Administration of "LodienT Tablet 80/2.5mg" and "TWYNSTA Tablet 80/5mg" in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety and PK of LODIENT Tablet 80/2.5mg in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HL-LDNT-101
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference (Active Comparator): TWYNSTA Tablet 80/5mg(Telmisartan/Amlodipine)
  Interventions: Drug: Twynsta
- Test (Experimental): LodienT Tablet 80/2.5mg(Telmisartan/S-amlodipine)
  Interventions: Drug: LodineT

INTERVENTIONS:
Drug: Twynsta — Manufactured by Boehringer Ingelheim
  Arms: Reference
Drug: LodineT — •Manufactured by Hanlim Pharm. Co., Ltd, Seoul, Korea
  Arms: Test

SUMMARY:
A randomized, open label, single dose, 2-sequence, 4-period, cross-over phase I clinical trial to compare and evaluate the safety and pharmacokinetics after oral administration of "LodienT tablet 80/2.5mg(telmisartan/s-amlodipine)" and "TWINSTA tablet 80/5mg(telmisartan/amlodipine)" in healthy adult volunteers.

DETAILED DESCRIPTION:
Amlodipine is a drug which belongs to calcium channel blockers (CCBs) and is used to treat hypertension. The molecule contains one chiral carbon atom and exists as a racemic mixture. As only the S-enantiomer of amlodipine [S-amlodipine] shows the CCB effect and R-amlodipine is responsible for the development of peripheral edema, purifying S-amlodipine can reduce the incidences of peripheral edema and other side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged more than 19 years old
2. Subject does not have congenital or chronic disease and is without pathologic symptom or finding on medical exam.
3. Subject was determined eligible according to the results of clinical laboratory tests like serum test, hematologic test, blood chemistry test, urine test etc. and vital signs, electrocardiography, physical exam etc. performed during the screening exam.
4. 90mmHg≤SBP≤139mmHg and 60mmHg≤DBP≤89mmHg)
5. Body mass index (BMI) of 18-30kg/m2
6. Willing and able to provide written informed consent

Exclusion Criteria:

1. Administration of other drug than can modulate metabolic enzyme within 1 months prior to the scrrening day.
2. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs
3. Continued excessive use of alcohol(alcohol>21 cups/day) and severe heavy smoker (cigarette > 20 cigarettes per day)
4. Administration of other investigational products within 6 months prior to the first dosing
5. Subject with the following conditions in laboratory test : AST(sGOT) or ALT(sGPT) > Upper normal limit × 1.5
6. Subject with whole blood donation within 60 days, component blood donation within 14 days, blood donation within 30 days
7. Subject who take a medication that affect to the pharmacokinetics of drug within 10 days
8. Subject with decision of non-participation through investigator's review

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-29 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
AUCt | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48 and 72hr
Cmax | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48 and 72hr

CONTACTS AND LOCATIONS:
Locations (1):
- Metro Hospital, Anyang, Kyung Gi, South Korea

IPD SHARING:
Plan to Share IPD: No